CLINICAL TRIAL: NCT05258305
Title: Prospective Study on Fat Retention When Using the AuraGen 1-2-3™ With AuraClens™ System in Processing of Lipoaspirate for Autologous Fat Grafting to the Breast
Brief Title: AuraClens™ System in Processing of Lipoaspirate for Autologous Fat Grafting to the Breast
Acronym: AuraGen
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tiger Biosciences, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AUG-002
Record Dates: First submitted 2022-02-17; First posted 2022-02-28 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Breast Fat Grafting Retention

STUDY DESIGN:
Intervention Model Description: This is a non-randomized open-label study with a patient population consisting of up to 200 subjects divided in 2 cohorts with 100 patients each: reconstruction and augmentation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Augmentation (Other): Subjects undergoing an aesthetic fat grafting procedure to the breast with or without a breast implant.
  Interventions: Device: AuraGen 1-2-3 with AuraClens
- Reconstruction (Other): Subjects undergoing reconstructive fat grafting procedure to the breast with or without a breast implant.
  Interventions: Device: AuraGen 1-2-3 with AuraClens

INTERVENTIONS:
Device: AuraGen 1-2-3 with AuraClens — Autologous fat transfer (AFT) is a minimally invasive medical procedure that includes aspirating adipose tissue from one part of the body, and washing, filtering and re-injecting the processed fat tissue into a different part of the body with the primary purpose of adding volume. The AuraGen 1-2-3 with AuraClens is a lipoaspirate wash system designed to be used in the operating room in conjunction with a user-provided liposuction cannular, a vacuum source, and waste canister.

SUMMARY:
Prospective, multi-center, non-randomized, open-label, post-market clinical study evaluating adipose graft retention over time from lipoaspirate processed using the AuraGen 1-2-3™ with AuraClens™ Lipoaspirate Wash System.

DETAILED DESCRIPTION:
Autologous fat transfer (AFT) is a medical procedure that includes aspirating adipose tissue from one part of the body, and washing, filtering and re-injecting the processed fat tissue into a different part of the body with the primary purpose of adding volume. The AuraGen1-2-3 with AuraClens Lipoaspirate Wash System is designed to be used in the operating room in conjunction with a user-provided liposuction cannular, a vacuum source, and waste canister. The study population will consist of up to 200 subjects in (2) cohorts: 100 subjects undergoing breast reconstruction and 100 subjects undergoing breast augmentation. All subjects will receive autologous lipoaspirate processed with the A123+ AuraClens and will be followed post-procedure at 1-, 3-, 6-, and 12-months. Fat graft retention will be evaluated with 3D imaging using the Canfield Vectra XT imaging system. Patient satisfaction will be measured between baseline and the post-procedure follow-up visits using a breast satisfaction questionnaire.

ELIGIBILITY:
Augmentation Subjects

Inclusion Criteria:

* Female patients > 22 years and < 65 years of age.
* Patients with a BMI < 35.
* Patients undergoing an aesthetic fat grafting procedure to the breast (breast augmentation) with or without a breast implant.
* Patients must be able to provide written informed consent, understand and be willing to comply with study-related procedures and follow-up visits.
* Patients must be non-smokers.
* Patients with available/adequate harvest sites for fat grafting.
* Anticipated harvested fat volume between 200 and 700 cc.
* Anticipated fat injection volume between 50 and 350 cc per breast.
* Anticipated breast implant volume between 200 and 550 cc.
* Patients must agree to maintain their weight (i.e., within 5%) by not making any major changes in diet or lifestyle during the study.

Exclusion Criteria:

* Skin rash in the treatment area.
* Patients who smoke or use nicotine products.
* Patients with bleeding disorders or currently taking anticoagulants.
* Patients with history of trauma or surgery to the treatment area.
* Patients with history of breast cancer.
* Active, chronic, or recurrent infection.
* Compromised immune system.
* Hypersensitivity to analgesic agents.
* Co-morbid condition that could limit ability to participate in the study or to comply with follow-up requirements.
* Untreated drug and/or alcohol abuse.
* Pregnant or breastfeeding.
* Any issue that, at the discretion of the Investigator, would contra-indicate the patient's participation.
* Patients who do not wish to have the study area (breast) photographed.

Reconstruction Subjects

Inclusion Criteria:

* Female patients > 18 years and < 65 years of age.
* Patients with a BMI < 35.
* Patients undergoing a fat grafting procedure to the breast in a second or third stage of a staged breast reconstruction, with or without a breast implant.
* Patient is at least 1 year post-completion of chemotherapy.
* Patients must be able to provide written informed consent, understand and be willing to comply with study-related procedures and follow-up visits.
* Patients must be non-smokers.
* Patients with available/adequate harvest sites for fat grafting.
* Anticipated harvested fat volume between 200 and 700 cc.
* Anticipated fat injection volume between 50 nd 350cc per breast.
* Anticipated breast implant volume (if applicable) between 200 and 550 cc.
* Patients must agree to maintain their weight (i.e., within 5%) by not making any major changes in diet or lifestyle during the study.

Exclusion Criteria:

* Skin rash in the treatment area.
* Patients who smoke or use nicotine products.
* Patients with bleeding disorders or currently taking anticoagulants.
* Patients undergoing active treatment for breast cancer.
* Active, chronic, or recurrent infection.
* Compromised immune system.
* Hypersensitivity to analgesic agents.
* Co-morbid condition that could limit ability to participate in the study or to comply with follow-up requirements.
* Untreated drug and/or alcohol abuse.
* Pregnant or breastfeeding.
* Any issue that, at the discretion of the Investigator, would contra-indicate the patient's participation.
* Patients who do not wish to have the study area (breast) photographed.

Ages: 22 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2022-05-05 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Fat Grafting Volume Retention | 1 Year
  Fat grafting volume retention change from baseline to 12-months.
Patient Satisfaction | 1 Year
  Sientra Breast Satisfaction Questionnaire survey results at 1, 3, 6 and 12-months post-operatively compared to baseline, based on a rating scale between 1 ("Strongly Disagree") to 7 ("Strongly Agree").

CONTACTS AND LOCATIONS:
Overall Officials: Denise Dajles, PhD, Study Director — Tiger Biosciences, LLC.
Locations (15):
- United States (15):
  - Tessler Plastic Surgery, Scottsdale, Arizona
  - Aura Aesthetica, Inc., Beverly Hills, California
  - Baptist Miami / Miami Cancer Institute, Miami, Florida
  - Meridian Plastic Surgery, Carmel, Indiana
  - Ascentist Plastic Surgery, Overland Park, Kansas
  - Calo Aesthetics, Louisville, Kentucky
  - Dallas Plastic Surgery, Metairie, Louisiana
  - V Plastic Surgery, West Long Branch, New Jersey
  - NYU Langone Plastic Surgery Associates, New York, New York
  - Luxurgery, New York, New York
  - Hunstad Kortesis Bharti Cosmetic Surgery, Huntersville, North Carolina
  - Restora Austin, Austin, Texas
  - Regional Plastic Surgery, Richardson, Texas
  - Dallas Plastic Surgery, University Park, Texas
  - Bellevue Plastic Surgery, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: No